CLINICAL TRIAL: NCT06146569
Title: Effects of Transcutaneous Vagus Nerve Stimulation (taVNS) in Individuals With Primary Dysmenorrhea: A Randomized Controlled Study
Brief Title: Effects of Transcutaneous Vagus Nerve Stimulation (taVNS) in Individuals With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vagus Nerve Stimulation
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dysmenorrhea Primary; Pain
Keywords: Dysmenorrhea; Menstrual cycle; Pain; Function
MeSH Terms: conditions — Pain; Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Two treatment groups have been formed to receive taVNS and sham taVNS.
Who Masked: Participant, Investigator
Masking Description: Throughout the study, participants and researchers involved in assessments and interventions will remain blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Auricular Vagus Nerve Stimulation (Experimental): Each patient in the Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) group will receive a treatment protocol consisting of taVNS. The treatment will be administered for five days beginning on the first day of pain experienced between the 1st and 2nd menstrual cycles.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
- Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham Comparator): Each patient in the sham Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) group will receive a treatment protocol consisting of sham taVNS. The treatment will be administered for five days beginning on the first day of pain experienced between the 1st and 2nd menstrual cycles.
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Current will be applied bilaterally from the tragus and turbinate parts of the ear with the VagustimTM device. The current frequency to be used in modulation mode is 10 Hz, and the pulse width is 300 μs (In modulation mode, the pulse rate and width are automatically changed in a loop pattern. The pulse width is reduced by 50% from its original setting in 0.5 seconds; then, the pulse rate is changed in 0.5 seconds, reduced by 50% from the original setting. Total cycle time is 1 second.). The current intensity will be applied for 5 minutes, keeping the current constant where the participant feels comfortable.
  Arms: Transcutaneous Auricular Vagus Nerve Stimulation
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — For 5 minutes, sham applications will be applied using a current-free headset specifically designed for this purpose. Participants will observe the device's functionality, but it will not supply any current.
  Arms: Sham Transcutaneous Auricular Vagus Nerve Stimulation

SUMMARY:
This study aims to investigate the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on pain, functional and emotional symptoms, and physical performance in individuals with primary dysmenorrhea (PD).

DETAILED DESCRIPTION:
In this study, which will be conducted over two menstrual cycles, 34 patients with PD will be randomised into two groups: taVNS and sham treatment. From the onset of pain during the menstrual cycle, taVNS or sham treatment will be applied for five days. Pain assessment will be conducted using the Numerical Rating Scale (NRS), pressure pain threshold with an algometer, menstrual symptoms using the Menstrual Symptom Scale (MSS) and the Functional and Emotional Measure of Dysmenorrhea (FEMD), anxiety using the Hamilton Anxiety Scale (HAM-A), and physical performance using the 6-Minute Walk Test (6MWT) during the first and second menstruation.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with PD according to the No. 345 Primary Dysmenorrhea Consensus Guidelines,
* An NRS score of at least three during menstruation before treatment,
* Being a woman between the ages of 18-40,
* A regular menstrual cycle of 28±7 days,
* Being nulliparous,
* No history of brain surgery, tumour or intracranial metal implantation,
* No chronic genitourinary infection or alcohol or drug use.

Exclusion Criteria:

* History of dizziness or epileptic disease,
* Pregnancy,
* Women with intrauterine devices,
* Metal implants in the head area,
* Women with skin lesions in the area where the electrodes will be placed,
* Use of analgesic drugs during treatment,
* Women with neurological or heart disease,
* Women are diagnosed with gynaecological conditions (endometriosis, adenomyosis, uterine fibroids, etc., which may be associated with secondary dysmenorrhea).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with primary dysmenorrhea will be included.
Enrollment: 50 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | On the 1st menstrual day before the intervention
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Intensity | On the 2nd menstrual day before the intervention
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Intensity | On the 3rd menstrual day before the intervention
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Intensity | On the 1st day of menstruation when the intervention occurred
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Intensity | On the 2nd day of menstruation when the intervention occurred
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Intensity | On the 3rd day of menstruation when the intervention occurred
  Numerical Rating Scale (NRS) data will be queried separately for lower abdominal, waist and bilateral thigh pain. Participants will be required to fill out an NRS questionnaire through the Google Forms web survey platform (Google LLC, Mountain View, CA, USA) before going to bed at night on days 1, 2, and 3 of two consecutive menstrual cycles. The questionnaire will be based on the most severe pain they experienced during the day. The minimum score of the NRS is 0, and the maximum score is 10. Higher scores are associated with more severe pain intensity.
Pain Pressure Threshold | On the 1st menstrual day before the intervention
  To measure the pressure pain threshold, it will be used a Push-Pull Force Gauge® (1200-304) will be used by Fabrication Enterprises, Inc. This handheld algometer allows linear force application ranging between 0 and 10 kg (22 lb × ¼ lb and 10 kg × 100 g). Initially, two exercises will be performed on the extensor muscles of the dominant forearm so that patients can become familiar with the equipment. The evaluator will position the algometer perpendicular to each point and apply gradual pressure at a constant rate of approximately 0.5 kg/cm2/s. The pressure will be increased until the participant reports feeling pain. Each point will be evaluated three times, and the average value will be recorded. The measurement will be performed on five reference points in the abdomen and one reference point in the lumbar spine, as in a previous study where pain was evaluated in PD.
Pain Pressure Threshold | Immediately after the intervention
  To measure the pressure pain threshold, it will be used a Push-Pull Force Gauge® (1200-304) will be used by Fabrication Enterprises, Inc. This handheld algometer allows linear force application ranging between 0 and 10 kg (22 lb × ¼ lb and 10 kg × 100 g). Initially, two exercises will be performed on the extensor muscles of the dominant forearm so that patients can become familiar with the equipment. The evaluator will position the algometer perpendicular to each point and apply gradual pressure at a constant rate of approximately 0.5 kg/cm2/s. The pressure will be increased until the participant reports feeling pain. Each point will be evaluated three times, and the average value will be recorded. The measurement will be performed on five reference points in the abdomen and one reference point in the lumbar spine, as in a previous study where pain was evaluated in PD.

SECONDARY OUTCOMES:
Menstrual Symptom Scale (MSS) | On the 1st menstrual day before the intervention
  The scale consists of 22 items and uses a 5-point Likert-type format. Participants are asked to rate the severity of their menstrual symptoms on a scale of 1 (never) to 5 (always). The scale contains three subscales: 'Negative Effects/Somatic Complaints' (items 1-13), 'Menstrual Pain Symptoms' (items 14-19), and 'Coping Methods' (items 20-22). The maximum score on the scale is 110, and the minimum score is 22. MSS score is calculated by taking the average score of all items in the scale. High scores are associated with increased menstrual symptoms.
Menstrual Symptom Scale (MSS) | Immediately after the intervention
  The scale consists of 22 items and uses a 5-point Likert-type format. Participants are asked to rate the severity of their menstrual symptoms on a scale of 1 (never) to 5 (always). The scale contains three subscales: 'Negative Effects/Somatic Complaints' (items 1-13), 'Menstrual Pain Symptoms' (items 14-19), and 'Coping Methods' (items 20-22). The maximum score on the scale is 110, and the minimum score is 22. MSS score is calculated by taking the average score of all items in the scale. High scores are associated with increased menstrual symptoms.
Functional and Emotional Measure of Dysmenorrhea (FEMD) | On the 1st menstrual day before the intervention
  Functional and Emotional Measure of Dysmenorrhea (FEMD), consisting of 14 items, evaluates dysmenorrhea functionally and emotionally with a 5-point Likert-type item. The reliability and validity study of the scale developed in 2012 was conducted in Turkey in 2015. As the scores obtained from the scale with a minimum score of 14 and a maximum score of 70 increase, the functional and emotional impact of dysmenorrhea also increases.
Functional and Emotional Measure of Dysmenorrhea (FEMD) | Immediately after the intervention
  Functional and Emotional Measure of Dysmenorrhea (FEMD), consisting of 14 items, evaluates dysmenorrhea functionally and emotionally with a 5-point Likert-type item. The reliability and validity study of the scale developed in 2012 was conducted in Turkey in 2015. As the scores obtained from the scale with a minimum score of 14 and a maximum score of 70 increase, the functional and emotional impact of dysmenorrhea also increases.
Hamilton Anxiety Scale (HAM-A) | On the 1st menstrual day before the intervention
  Patients with chronic pain often experience mood disorders, such as depression and anxiety. The Hamilton Anxiety Scale (HAM-A) will be used to assess the intensity of anxiety symptoms. The scale measures both mental and physical anxiety with 14 symptom-defined items. Each item is scored from 0 (not present) to 4 (severe). The total score range is 0-56. On the anxiety scale, scores of 17 or below indicate mild anxiety, while scores of 18-24 indicate moderate anxiety, and scores of 25-30 indicate severe anxiety.
Hamilton Anxiety Scale (HAM-A) | Immediately after the intervention
  Patients with chronic pain often experience mood disorders, such as depression and anxiety. The Hamilton Anxiety Scale (HAM-A) will be used to assess the intensity of anxiety symptoms. The scale measures both mental and physical anxiety with 14 symptom-defined items. Each item is scored from 0 (not present) to 4 (severe). The total score range is 0-56. On the anxiety scale, scores of 17 or below indicate mild anxiety, while scores of 18-24 indicate moderate anxiety, and scores of 25-30 indicate severe anxiety.
6-Minute Walk Test (6MWT) | On the 1st menstrual day before the intervention
  The 6-Minute Walk Test (6MWT) will evaluate submaximal functional capacity. 6MWT measures the maximum distance participants can walk as quickly as possible for 6 minutes.
6-Minute Walk Test (6MWT) | Immediately after the intervention
  The 6-Minute Walk Test (6MWT) will evaluate submaximal functional capacity. 6MWT measures the maximum distance participants can walk as quickly as possible for 6 minutes.
Positive and Negative Affect Schedule (PANAS) | On the 1st menstrual day before the intervention
  For taVNS administration, the positive and negative affect will be assessed before and after treatment using the Positive and Negative Affect Schedule (PANAS). This 5-point Likert-type scale was developed in 1988 and includes 20 items: 10 positive and 10 negative. A score range of 10-50 assesses both positive and negative effects.
Positive and Negative Affect Schedule (PANAS) | Immediately after the intervention
  For taVNS administration, the positive and negative affect will be assessed before and after treatment using the Positive and Negative Affect Schedule (PANAS). This 5-point Likert-type scale was developed in 1988 and includes 20 items: 10 positive and 10 negative. A score range of 10-50 assesses both positive and negative effects.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Lecturer, Principal Investigator — Artvin Coruh University
Locations (1):
- Zeynep Yıldız Kızkın, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burnett M, Lemyre M. No. 345-Primary Dysmenorrhea Consensus Guideline. J Obstet Gynaecol Can. 2017 Jul;39(7):585-595. doi: 10.1016/j.jogc.2016.12.023. PMID 28625286
- [Background] Itani R, Soubra L, Karout S, Rahme D, Karout L, Khojah HMJ. Primary Dysmenorrhea: Pathophysiology, Diagnosis, and Treatment Updates. Korean J Fam Med. 2022 Mar;43(2):101-108. doi: 10.4082/kjfm.21.0103. Epub 2022 Mar 17. PMID 35320895
- [Background] Karout S, Soubra L, Rahme D, Karout L, Khojah HMJ, Itani R. Prevalence, risk factors, and management practices of primary dysmenorrhea among young females. BMC Womens Health. 2021 Nov 8;21(1):392. doi: 10.1186/s12905-021-01532-w. PMID 34749716
- [Background] Ju H, Jones M, Mishra G. The prevalence and risk factors of dysmenorrhea. Epidemiol Rev. 2014;36:104-13. doi: 10.1093/epirev/mxt009. Epub 2013 Nov 26. PMID 24284871
- [Background] Habibi N, Huang MS, Gan WY, Zulida R, Safavi SM. Prevalence of Primary Dysmenorrhea and Factors Associated with Its Intensity Among Undergraduate Students: A Cross-Sectional Study. Pain Manag Nurs. 2015 Dec;16(6):855-61. doi: 10.1016/j.pmn.2015.07.001. Epub 2015 Aug 29. PMID 26328887
- [Background] Wang L, Wang Y, Wang Y, Wang F, Zhang J, Li S, Wu M, Li L, Rong P. Transcutaneous auricular vagus nerve stimulators: a review of past, present, and future devices. Expert Rev Med Devices. 2022 Jan;19(1):43-61. doi: 10.1080/17434440.2022.2020095. Epub 2022 Jan 13. PMID 34937487
- [Background] Wang YJ, Hsu CC, Yeh ML, Lin JG. Auricular acupressure to improve menstrual pain and menstrual distress and heart rate variability for primary dysmenorrhea in youth with stress. Evid Based Complement Alternat Med. 2013;2013:138537. doi: 10.1155/2013/138537. Epub 2013 Dec 12. PMID 24416063
- [Background] Pegado R, Silva LK, da Silva Dantas H, Andrade Camara H, Andrade Mescouto K, Silva-Filho EM, Lopes JM, Micussi MTABC, Correia GN. Effects of Transcranial Direct Current Stimulation for Treatment of Primary Dysmenorrhea: Preliminary Results of a Randomized Sham-Controlled Trial. Pain Med. 2020 Dec 25;21(12):3615-3623. doi: 10.1093/pm/pnz202. PMID 31498389
- [Background] Dutra LRDV, Pegado R, Silva LK, da Silva Dantas H, Camara HA, Silva-Filho EM, Correia GN, Micussi MTABC. Modulating Anxiety and Functional Capacity with Anodal tDCS Over the Left Dorsolateral Prefrontal Cortex in Primary Dysmenorrhea. Int J Womens Health. 2020 Apr 5;12:243-251. doi: 10.2147/IJWH.S226501. eCollection 2020. PMID 32308497
- [Background] Kane RL, Bershadsky B, Rockwood T, Saleh K, Islam NC. Visual Analog Scale pain reporting was standardized. J Clin Epidemiol. 2005 Jun;58(6):618-23. doi: 10.1016/j.jclinepi.2004.11.017. PMID 15878476
- [Derived] Yildiz Kizkin Z, Yildiz R, Ozden AV. Effects of Transcutaneous Auricular Vagus Nerve Stimulation in Individuals with Primary Dysmenorrhea: A Randomized Controlled Trial. Neuromodulation. 2025 Oct 17:S1094-7159(25)01031-1. doi: 10.1016/j.neurom.2025.09.306. Online ahead of print. PMID 41108303

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06146569/Prot_SAP_000.pdf